CLINICAL TRIAL: NCT01560221
Title: Reducing Drug Use and HIV Risk in Drug-dependent Adults Arrested for Prostitution
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Anthony DeFulio, Assistant Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R34DA033141 (NIH)
Record Dates: First submitted 2012-03-15; First posted 2012-03-22 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Substance-related Disorders; HIV Risk Behavior
MeSH Terms: conditions — Substance-Related Disorders | interventions — Methadone; Buprenorphine; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Therapeutic Workplace (Experimental): Participants will receive all standard services plus the Therapeutic Workplace intervention, in which access to stipend supported training and/or wage subsidies for community employment is contingent upon drug abstinence as verified by urinalysis.
  Interventions: Behavioral: Therapeutic Workplace; Drug: Methadone; Drug: Buprenorphine
- Standard Services (Active Comparator): Participants will receive methadone treatment or buprenorphine treatment, depending upon medical recommendations of their physicians, slot availability, and their own preferences. Participants who remain in treatment for at least 90 days will have the charge of prostitution that is pending against them dropped.
  Interventions: Drug: Methadone; Drug: Buprenorphine

INTERVENTIONS:
Behavioral: Therapeutic Workplace — Participants can access stipend supported academic and job skills training for adults and/or receive wages or wage subsides for actual employment. Access to training and employment is contingent upon meeting therapeutic targets. Potential targets include, but are not limited to, drug abstinence and medication adherence.
  Arms: Therapeutic Workplace
Drug: Methadone — Methadone in liquid form, with the dosage determined by physician on an individual basis. Anticipated dose range 30mg to 100mg daily. Methadone is administered daily at a methadone clinic for as long as enrollment in the methadone clinic is maintained.
Drug: Buprenorphine — Subutex (buprenorphine hydrochloride) and Suboxone tablets (buprenorphine hydrochloride and naloxone hydrochloride) are approved for the treatment of opiate dependence. Subutex and Suboxone treat opiate addiction by preventing symptoms of withdrawal from heroin and other opiates.
  Other Names: Suboxone, Subutex

SUMMARY:
The combination of using injection drugs, smoking crack cocaine, having multiple sex partners, and inconsistent condom use results in substantial risk for acquiring and transmitting HIV, and many drug dependent adults who have been arrested on charges of prostitution fit this profile. Existing interventions for reducing HIV risk have had limited efficacy in drug-dependent sex workers, and criminal justice approaches have been ineffective despite their high cost. A potentially ideal alternative is to divert drug-dependent arrestees from prosecution to a treatment that reduces drug use and HIV sex risk behaviors, while providing job skills training and promoting community employment to alleviate the financial need to continue sex work. In order to provide an effective therapeutic alternative to criminal prosecution, the investigators propose to develop a multifaceted intervention that includes opiate agonist treatment (i.e., methadone OR buprenorphine) and the Therapeutic Workplace. The Therapeutic Workplace is a supported environment in which participants are required to provide drug-free urine samples to access paid job skills training or employment and to maintain the maximum rate of pay. The overall intervention is designed to reduce drug use and HIV risk behaviors, and simultaneously promote employment. The proposed project is a 2-year Stage I behavior therapy development effort that will include the development, manualization and pilot testing of a Therapeutic Workplace intervention tailored to drug-dependent adults arrested for prostitution. In the pilot study, the investigators will recruit opiate- and cocaine-dependent adults arrested for prostitution from the Eastside District Court in Baltimore. Eligible individuals will be offered methadone treatment in lieu of prosecution and will be required to remain in methadone treatment for 90 days to have the charges against them dropped. After enrolling in opiate agonist treatment, the diverted individuals will be invited to participate in the pilot study. Interested individuals will be randomly assigned to receive the standard opiate agonist treatment services or these services plus the Therapeutic Workplace. The Therapeutic Workplace has two phases. In Phase 1, participants will be offered four months of stipend-supported job training in the Therapeutic Workplace. In Phase 2, participants will be encouraged to seek employment in a community job and will receive wage subsidies for four months for maintaining community employment or engaging in supervised job seeking. Throughout both phases, participants will be required to provide drug-free urine samples to receive Therapeutic Workplace wages (training stipends in Phase 1 and wage subsidies in Phase 2). The wage subsidy program will include drug testing managed by a national supplier of drug-free workplace services. Overall, this treatment could serve as a novel and ideal intervention for drug-dependent adults arrested for prostitution while reducing criminal justice costs.

ELIGIBILITY:
Inclusion criteria:

* Opioid dependent
* Adults
* Recently arrested
* Have a pending charge of prostitution or perverted practice

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Drug abstinence | Participants will be followed for eight months. Drug abstinence will be measured every 30 days throughout the eight month period.
  A combination of urinalysis and self-reports of illicit drug use. This outcome is treated as dichotomous: Urine samples are considered positive or negative based on standard cutoffs for drugs of abuse, and self-reports are yes or no depending upon whether there was or was not any drug use in the previous 30 days.

SECONDARY OUTCOMES:
HIV Sex Risk | Participants will be followed for eight months. HIV Sex Risk will be measured every 30 days throughout the eight month period.
  The self-reported number of unprotected vaginal and anal sex occasions in the prior month.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony DeFulio, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- The Center for Learning and Health, Baltimore, Maryland, United States